CLINICAL TRIAL: NCT00317707
Title: Risk and Prevention Study: Optimisation of the Preventive Strategies and Evaluation of the Efficacy of n-3 PUFA in Subjects at High Cardiovascular Risk
Brief Title: Risk and Prevention Study: Evaluation of the Efficacy of n-3 PUFA in Subjects at High Cardiovascular Risk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R&P
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular risk; cardiovascular diseases; cardiovascular prevention; polyunsaturated fatty acids; diabetes; hypertension; hypercholesterolemia; obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Obesity | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-3 PUFA (Experimental)
  Interventions: Drug: N-3 Polyunsaturated Fatty Acids
- Olive oil (Placebo Comparator)
  Interventions: Drug: Placebo: Olive oil

INTERVENTIONS:
Drug: N-3 Polyunsaturated Fatty Acids — Each subject assigned to active treatment group will receive 1g/day capsule of n-3 PUFA
  Arms: N-3 PUFA
Drug: Placebo: Olive oil — Each subject assigned to the control group will receive 1 g/day capsule of olive oil.
  Arms: Olive oil

SUMMARY:
In the everyday practice cardiovascular prevention in people at high risk is still unsatisfactory and treatments with documented efficacy are generally under-used.

Polyunsaturated fatty acids of marine origin (n-3 PUFA) are the latest more promising strategy to improve prognosis in these patients.

The Risk and Prevention study combines an epidemiological and an experimental approach in order to:

1. Verify the possibility to optimise cardiovascular prevention in subjects at high risk by planning the intervention with patients and setting individual goals (outcome study)
2. Evaluate the efficacy of a long term n-3 PUFA treatment in reducing the incidence of cardiovascular events, through a controlled, randomised, double blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Multiple risk factors:

  * diabetes,
  * age => 65 years,
  * male sex,
  * hypertension,
  * hypercholesterolemia,
  * smoking,
  * obesity,
  * family history of premature cardiovascular disease;
* Previous manifestations of atherosclerotic disease (ischemic stoke, transient ischemic attack [TIA], peripheral artery disease, previous arterial revascularisation procedures, angina pectoris)

Exclusion Criteria:

* Contraindications (known allergies to n-3 PUFA) or indications (previous myocardial infarction) for the treatment with n-3 PUFA
* Serious comorbidity with an unfavourable prognosis over the short term
* Expected non compliance over a long period of time
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12513 (Actual)
Dates: Start 2004-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
cardiovascular deaths and hospitalization for cardiovascular causes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tombesi Massimo, MD, Study Chair — Centro Studi e Ricerca in Medicina Generale, Monza, Italy; Tognoni Gianni, MD, Study Chair — Mario Negri Institute for Pharmacological Research, Milan, Italy
Locations (1):
- Mario Negri Institute for Pharmacological Research, Milan, Italy

REFERENCES:
- [Derived] Risk and Prevention Study Collaborative Group; Roncaglioni MC, Tombesi M, Avanzini F, Barlera S, Caimi V, Longoni P, Marzona I, Milani V, Silletta MG, Tognoni G, Marchioli R. n-3 fatty acids in patients with multiple cardiovascular risk factors. N Engl J Med. 2013 May 9;368(19):1800-8. doi: 10.1056/NEJMoa1205409. PMID 23656645
- [Derived] Rischio and Prevenzione Investigators. Efficacy of n-3 polyunsaturated fatty acids and feasibility of optimizing preventive strategies in patients at high cardiovascular risk: rationale, design and baseline characteristics of the Rischio and Prevenzione study, a large randomised trial in general practice. Trials. 2010 May 28;11:68. doi: 10.1186/1745-6215-11-68. PMID 20509875